CLINICAL TRIAL: NCT03867942
Title: Randomized, Open-label, Single Dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics/Pharmacodynamics, Safety, and Tolerability of the Monolayer Drug in Comparison to the Bilayer Drug Administered in Healthy Volunteers
Brief Title: BE Study of Bilayer Combination of Gemigliptin/Rosuvastatin 50/20mg in Comparison to Monolayer Combination.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-GSCL006
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2; Dyslipidemias
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monolayer group (Active Comparator): monolayer of Gemigliptin/Rosuvastatin
  Interventions: Drug: Monolayer group; Drug: Bilayer group
- bilayer group (Experimental): bilayer of Gemigliptin/Rosuvastatin
  Interventions: Drug: Monolayer group; Drug: Bilayer group

INTERVENTIONS:
Drug: Monolayer group — Monolayered combination of gemigliptin and rosuvastatin
Drug: Bilayer group — Bilayered combination of gemigliptin and rosuvastatin

SUMMARY:
To evaluate and compare PK/PD, safety and tolerability of monolayer combination of Gemigliptin/Rosuvastatin 50/20mg and bilayer combination of Gemigliprin/Rosuvastatin 50/20mg in healthy adults.

DETAILED DESCRIPTION:
To evaluate and compare Pharmacokinetics/Pharmacodynamics, safety and tolerability of monolayer combination of Gemigliptin/Rosuvastatin 50/20mg in comparison to bilayer combination of Gemigliprin/Rosuvastatin 50/20mg administered in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age: 19~45
* Body weight: 55kg or higher(female: 50kg or higher) and BMI 18~27kg/m2
* SBP 90~150mmHg, DBP 60-95mmHg
* Fasting glucose 70~120mg/dL
* Infertility

  1. Surgically infertile
  2. To prevent pregnancy, participants who agreed using 2 or more contraceptive methods. Such as
* Barrier methods: Condom, Diaphragm, Cervical cap (Pessary), Spermicide
* Hormonal methods: Pills, Injection (Depot), Skin patch, Hormonal implant (Implanon), Vaginal ring
* Intrauterine Devices (IUDs): Cooper IUD (Loop), Hormonal IUD (Mirena)
* Natural methods: Basic body temperature, Ovulation period, Coitus interruptus, Abstinent
* People who perfectly understood clinical trial and independently decided to participate in clinical trial.
* People who will be able to collect blood sample during clinical trial period.
* People who are suitable to participate clinical trial by physical examination, lab test and medical examination by interview.

Exclusion Criteria:

* Genetic problems such as galactose intolerance, Lapp lacatase deficiency, glucose-galactose malabsorption
* Clinically significant disease such as liver, kidney, digestive, pulmonary, endocrine system, cardiovascular disease etc.
* People who have gastrointestinal disease or history of surgery which would affect absorption of drug.
* History of clinically significant drug induced hyper-sensitive reaction or drug related muscular disease

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-03-21 (Estimated); Primary Completion 2019-05-24 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Gemigliptin AUC | 0hour(pre-dose), 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 5hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour
  Gemigliptin
Rosuvastain AUC | 0hour(pre-dose), 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 5hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour
  Rosuvastain
Rosuvastain Cmax | 0hour(pre-dose), 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 5hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour
  Rosuvastain
Gemigliptin Cmax | 0hour(pre-dose), 0.5hour, 1hour, 1.5hour, 2hour, 3hour, 4hour, 5hour, 6hour, 8hour, 12hour, 24hour, 48hour, 72hour
  Gemigliptin

CONTACTS AND LOCATIONS:
Overall Officials: kyungsang Yoo, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No